CLINICAL TRIAL: NCT06008704
Title: Pathophysiology of Pain in Parkinson's Disease: Exploration of the Serotonin System in Positron Emission Tomography (PET [18F]-MPPF)
Brief Title: Pain in Parkinson's Disease: Exploration of the Serotonin System in Positron Emission Tomography (PET [18F]-MPPF)
Acronym: PD-Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/21/0566; 2022-501123-24 (EudraCT Number)
Record Dates: First submitted 2023-05-10; First posted 2023-08-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: PD-related central pain; PET [18F] MPPF; serotoninergic system; multimodal imaging; pain threshold
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: physio-pathological prospective open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients with central chronic pain (Other): Patients from both groups will receive the same interventions, the difference between groups is the eligibility criteria. In this arm only patients presenting central chronic pain will be included
  Interventions: Diagnostic Test: Clinical assessment; Diagnostic Test: Pain characteristics assessment; Diagnostic Test: MRI; Diagnostic Test: Thermotest; Diagnostic Test: UPDRS-III Scale; Diagnostic Test: [18F]-MPPF PET scan
- PD patients without pain (Other): Patients from both groups will receive the same interventions, the difference between groups is the eligibility criteria. In this arm only patients without central chronic pain will be included
  Interventions: Diagnostic Test: Clinical assessment; Diagnostic Test: Pain characteristics assessment; Diagnostic Test: MRI; Diagnostic Test: Thermotest; Diagnostic Test: UPDRS-III Scale; Diagnostic Test: [18F]-MPPF PET scan

INTERVENTIONS:
Diagnostic Test: Clinical assessment — The clinical assessment consists on behavioural and motor evaluations to determine the characteristics of the population
Diagnostic Test: Pain characteristics assessment — The pain characteristics assessment will be made with a variety of scales and questionnaires which allow to identify the extent of central pain and functional impairment
Diagnostic Test: MRI — The MRI examination allows anatomical imaging, diffusion imaging and functional imaging to measure specific markers
Diagnostic Test: Thermotest — The thermotest is performed to assess the pain perception threshold
Diagnostic Test: UPDRS-III Scale — The UPDRS-III scale allows to asses motor functionality of PD patients
Diagnostic Test: [18F]-MPPF PET scan — The PET scan after injection of [18F]-MPPF at a dose of 200 Megabecquerel/kg +/-10% allows in vivo imaging of 5HT1A receptors

SUMMARY:
This project will explore the involvement of the serotonin system in the pathophysiology of PD-related central pain. Thus, the serotonin system will be evaluated in PD patients with and without central pain who will benefit from brain positron emission tomography (PET) allowing in vivo imaging of 5HT1A receptors and multimodal brain MRI including morphometric imaging and functional connectivity (resting state acquisition).

DETAILED DESCRIPTION:
The prevalence of chronic pain in PD can be estimated at 60-80% from several epidemiological studies. Both semiological and pathophysiological classification proposes specific and non-specific pain in PD. While non-specific pain is not directly related to PD but may be aggravated by the disease, specific pain is a direct result of the disease with dystonic pain characterized by painful cramps in relation to motor symptoms and non-systematic central pain such as burning, paresthesia, compression (central parkinsonian pain). A case-control study reported that cramp-like pain and central pain were three times more frequent in parkinsonian patients than in the general population. Pathophysiologically, several studies suggest an abnormal nociceptive integration process in PD patients. Previous studies have indicated that the nociceptive signal is amplified along the pain transmission pathways. This could be related to increased facilitation through central sensitization of pain pathways or decreased inhibition (reduced activity of descending inhibitory control systems). Several recent studies suggest that the noradrenergic and/or serotonergic systems may be involved in the pathophysiology of PD-related pain. Therefore, this project will explore the involvement of the serotonergic system in the pathophysiology of pain using brain neuroimaging in PD patients with central pain.

The present study hypothesize that the binding of the radiotracer [18F]-MPPF, allowing in vivo imaging of 5HT1A receptors, will be reduced in PD patients with central pain compared to non-painful PD patients at the level of the median raphe, but also at the level of several brain structures involved in the pain matrix such as the insula, the anterior and posterior cingulate cortex, the orbitofrontal cortex, etc. A correlation between the clinical parameters of pain and the brain structures in which MRP binding is decreased should make it possible to confirm the link between these serotonin binding anomalies and pain. Finally, the morphological and functional MRI study should make it possible to identify structural and functional abnormalities within the pain networks in painful Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD defined according to United Kingdom Parkinson's Disease Brain Bank (UKPDSBB) criteria
* Patients with stable anti-parkinsonian treatment for at least 4 weeks prior to inclusion
* Patients with a Montreal Cognitive Assessment (MoCA) score > 25
* Patients with a Hospital Anxiety and Depression Scale (HADS)-D score ≥ 11
* Person affiliated or benefiting from a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

  • For patients with pain
* Patients with PD-related central pain defined according to the criteria of Marques et al, 2019
* Patients with chronic central pain (i.e. present for at least 3 months)
* Patients who have average pain over the previous month according to a VAS ≥ 4.

  • For patients without pain
* Patients who do not have pain defined as VAS ≤ 4, meaning that it does not interfere with daily activity.

Exclusion Criteria:

* Patients treated with second line therapy
* Patients with a history of significant psychiatric pathology according to the investigator
* Patients treated with drugs interacting with 5HT1A receptors in the previous 4 weeks
* Patients with contraindication to MRI
* Patients refusing to be informed of an abnormality discovered during brain imaging
* Patients with dyskinesias judged by the investigator to be disabling for imaging.
* Patients under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision
* Pregnant woman, breastfeeding woman

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Distribution volume ratio of [18F]-MPPF | during the procedure
  The MRP [18F]-MPPF marking the 5 HT1A receptors allows the in vivo visualization of serotonergic neurons and it's sensitive to extracellular variations of serotonin

SECONDARY OUTCOMES:
Pain intensity and [18F]-MPPF uptake | during the procedure
  Correlation between [18F]-MPPF uptake and central pain intensity measured with the Visual Analog Score for pain (Scale from 0 to 10, 10 being the most fote intensity of pain)
Functional impairment and [18F]-MPPF uptake | during the procedure
  Correlation between [18F]-MPPF uptake and functional impairment, measured with the Primary Parkinsonian Pain Diagnostic Questionnaire .
  It is a 39-item self-questionnaire evaluating the motor and psychological quality of life of Parkinson's patients over the past month. Each question is rated from 0 (no disturbance) to 4 (maximum disturbance), and items are divided into 8 dimensions (mobility, activities of daily life, emotional well-being, psychological discomfort, social support, cognitive disorders, communication, physical discomfort).
  A score is calculte in percentage. The higher the score, the lower the quality of life in this dimension. It is a simple and fast scale of transfer, reliable and validated, sensitive to change.
Pain perception thresholds and [18F]-MPPF uptake | during the procedure
  Correlation between [18F]-MPPF uptake and pain perception thresholds, measured with the thermotest
Macrostructural markers | during the procedure
  Measurement of macrostructural markers obtained by MRI Macrostructural markers measured by T1 and T2 sequences: density of gray matter
Central pain characteristics measured by Visual Analog Score for pain (VAS) and brain macrostructural markers | during the procedure
  Correlation between brain macrostructural markers and central pain characteristics measured with the Visual Analog Score for pain (VAS) which consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
5HT1A-receptors specific radioligand binding and functional networks connectivity | during the procedure
  Correlation between 5HT1A receptors specific radioligand binding and functional networks connectivity, obtained by IRM
Behavioral population characteristics obtained with the Hospital Anxiety and Depression scale (HAD) | during the procedure
  Mean of patient's behavioral characteristics score obtained with the Hospital Anxiety and Depression scale (HAD) which is scored between 0 meaning no impairment and 3 being severe impairment
Motor population characteristics obtained with the Movement Disorders Society-sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | during the procedure
  Mean of patient's motor characteristics score obtained with the Movement Disorders Society-sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS), which score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL-COURBON, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Centre Hospitalier Universitaire de Toulouse, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aznavour N, Zimmer L. [18F]MPPF as a tool for the in vivo imaging of 5-HT1A receptors in animal and human brain. Neuropharmacology. 2007 Mar;52(3):695-707. doi: 10.1016/j.neuropharm.2006.09.023. Epub 2006 Nov 13. PMID 17101155
- [Background] Boussac M, Arbus C, Dupouy J, Harroch E, Rousseau V, Ory-Magne F, Rascol O, Moreau C, Maltete D, Rouaud T, Meyer M, Houvenaghel JF, Marse C, Tranchant C, Hainque E, Jarraya B, Ansquer S, Bonnet M, Belamri L, Tir M, Marques AR, Danaila T, Eusebio A, Devos D, Brefel-Courbon C; PREDI-STIM study group*. Personality Dimensions Are Associated with Quality of Life in Fluctuating Parkinson's Disease Patients (PSYCHO-STIM). J Parkinsons Dis. 2020;10(3):1057-1066. doi: 10.3233/JPD-191903. PMID 32444557
- [Background] Boussac M, Arbus C, Dupouy J, Harroch E, Rousseau V, Croiset A, Ory-Magne F, Rascol O, Moreau C, Rolland AS, Maltete D, Rouaud T, Meyer M, Drapier S, Giordana B, Anheim M, Hainque E, Jarraya B, Benatru I, Auzou N, Belamri L, Tir M, Marques AR, Thobois S, Eusebio A, Corvol JC, Devos D, Brefel-Courbon C; PREDI-STIM study group. Personality dimensions of patients can change during the course of parkinson's disease. PLoS One. 2021 Jan 7;16(1):e0245142. doi: 10.1371/journal.pone.0245142. eCollection 2021. PMID 33411732
- [Background] Boussac M, Arbus C, Klinger H, Eusebio A, Hainque E, Corvol JC, Rascol O, Rousseau V, Harroch E, d'Apollonia CS, Croiset A, Ory-Magne F, De Barros A, Fabbri M, Moreau C, Rolland AS, Benatru I, Anheim M, Marques AR, Maltete D, Drapier S, Jarraya B, Hubsch C, Guehl D, Meyer M, Rouaud T, Giordana B, Tir M, Devos D, Brefel-Courbon C; PREDISTIM study group. Personality Related to Quality-of-Life Improvement After Deep Brain Stimulation in Parkinson's Disease (PSYCHO-STIM II). J Parkinsons Dis. 2022;12(2):699-711. doi: 10.3233/JPD-212883. PMID 34897100
- [Background] Brefel-Courbon C, Grolleau S, Thalamas C, Bourrel R, Allaria-Lapierre V, Loi R, Micallef-Roll J, Lapeyre-Mestre M. Comparison of chronic analgesic drugs prevalence in Parkinson's disease, other chronic diseases and the general population. Pain. 2009 Jan;141(1-2):14-8. doi: 10.1016/j.pain.2008.04.026. Epub 2008 Dec 4. PMID 19062167
- [Background] Brefel-Courbon C, Ory-Magne F, Thalamas C, Payoux P, Rascol O. Nociceptive brain activation in patients with neuropathic pain related to Parkinson's disease. Parkinsonism Relat Disord. 2013 May;19(5):548-52. doi: 10.1016/j.parkreldis.2013.02.003. Epub 2013 Feb 23. PMID 23462484
- [Background] Brefel-Courbon C, Payoux P, Thalamas C, Ory F, Quelven I, Chollet F, Montastruc JL, Rascol O. Effect of levodopa on pain threshold in Parkinson's disease: a clinical and positron emission tomography study. Mov Disord. 2005 Dec;20(12):1557-63. doi: 10.1002/mds.20629. PMID 16078219
- [Background] Chaudhuri KR, Schapira AH. Non-motor symptoms of Parkinson's disease: dopaminergic pathophysiology and treatment. Lancet Neurol. 2009 May;8(5):464-74. doi: 10.1016/S1474-4422(09)70068-7. PMID 19375664
- [Background] Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group. King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation. Mov Disord. 2015 Oct;30(12):1623-31. doi: 10.1002/mds.26270. Epub 2015 Jun 11. PMID 26096067
- [Background] Cloninger CR. Temperament and personality. Curr Opin Neurobiol. 1994 Apr;4(2):266-73. doi: 10.1016/0959-4388(94)90083-3. PMID 8038587
- [Background] Costes N, Merlet I, Zimmer L, Lavenne F, Cinotti L, Delforge J, Luxen A, Pujol JF, Le Bars D. Modeling [18 F]MPPF positron emission tomography kinetics for the determination of 5-hydroxytryptamine(1A) receptor concentration with multiinjection. J Cereb Blood Flow Metab. 2002 Jun;22(6):753-65. doi: 10.1097/00004647-200206000-00014. PMID 12045674
- [Background] Dellapina E, Gerdelat-Mas A, Ory-Magne F, Pourcel L, Galitzky M, Calvas F, Simonetta-Moreau M, Thalamas C, Payoux P, Brefel-Courbon C. Apomorphine effect on pain threshold in Parkinson's disease: a clinical and positron emission tomography study. Mov Disord. 2011 Jan;26(1):153-7. doi: 10.1002/mds.23406. Epub 2010 Oct 19. PMID 20960436
- [Background] Dellapina E, Pellaprat J, Adel D, Llido J, Harroch E, Martini JB, Kas A, Salabert AS, Ory-Magne F, Payoux P, Brefel-Courbon C. Dopaminergic denervation using [123I]-FPCIT and pain in Parkinson's disease: a correlation study. J Neural Transm (Vienna). 2019 Mar;126(3):279-287. doi: 10.1007/s00702-019-01974-5. Epub 2019 Jan 31. PMID 30706197
- [Background] Defazio G, Berardelli A, Fabbrini G, Martino D, Fincati E, Fiaschi A, Moretto G, Abbruzzese G, Marchese R, Bonuccelli U, Del Dotto P, Barone P, De Vivo E, Albanese A, Antonini A, Canesi M, Lopiano L, Zibetti M, Nappi G, Martignoni E, Lamberti P, Tinazzi M. Pain as a nonmotor symptom of Parkinson disease: evidence from a case-control study. Arch Neurol. 2008 Sep;65(9):1191-4. doi: 10.1001/archneurol.2008.2. PMID 18779422